CLINICAL TRIAL: NCT00761410
Title: A Prospective, Non-Comparative Multi Centre Study to Evaluate the Clinical Performance of the DePuy Press Fit Condylar (P.F.C.) Sigma Rotating Platform High Flexion Knee.
Brief Title: A Study to Determine the Performance of the Press Fit Condylar (P.F.C.) Sigma RP-F Knee System
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was terminated early due to prolonged recruitment period.
Sponsor: DePuy International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT0153
Record Dates: First submitted 2008-09-26; First posted 2008-09-29 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2016-06

CONDITIONS: Osteoarthritis
Keywords: Arthroplasty; Knee; Replacement; High Flexion; PFC Sigma RP-F
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- P.F.C. Sigma RP-F Total Knee Replacement (Other): An orthopaedic implant for total knee replacement with a mobile-bearing and a high flexion design
  Interventions: Device: P.F.C. Sigma RP-F Total Knee Replacement

INTERVENTIONS:
Device: P.F.C. Sigma RP-F Total Knee Replacement — An orthopaedic implant for total knee replacement with a mobile-bearing and a high flexion design

SUMMARY:
The purpose of this study is to evaluate if the P.F.C. Sigma RPF knee accommodates functional stability with a post-operative passive range of motion of greater than 125° of flexion and to demonstrate that the range of motion does not compromise the longevity of the implant.

DETAILED DESCRIPTION:
Primary endpoint is to demonstrate that 90% of patients have a functionally stable knee that can achieve post operative range of motion of 125 degrees or greater.

The secondary endpoint is to investigate the survivorship of the P.F.C. Sigma RP-F knee at 1, 2, 3, 5, 10, 15 and 20 years

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, aged between 45 and 75 years inclusive.
* Subjects who are able to give voluntary, written informed consent to participate in this investigation and from whom consent has been obtained.
* Subjects who are able to achieve a pre-operative passive range of motion of equal to or greater than 110º.
* Subjects who, in the opinion of the Investigator, are able to understand this investigation, co-operate with the investigational procedures and are willing to return to the hospital for all the required post-operative follow-ups.
* Subjects who present with idiopathic osteoarthritis that in the opinion of the clinical investigator requires a primary total knee arthroplasty.
* Subjects who in the opinion of the Clinical Investigator are considered to be suitable for treatment with the P.F.C.® Sigma RPF knee, according to the indications specified in the package insert leaflet.

Exclusion Criteria:

* Subjects who, in the opinion of the Investigator, have an existing condition that would compromise their participation and follow-up in this study.
* Women who are pregnant.
* Subjects who are known drug or alcohol abusers or with psychological disorders that could effect follow-up care or treatment outcomes.
* Subjects who have participated in a clinical study with an investigational product in the last month (30 days).
* Subjects who are currently involved in any personal injury litigation claims.
* Subjects with a known history of poor compliance to medical treatment.
* Subjects who have a pre-operative limb deformity of equal to or greater than 10° varus or 15° valgus as defined using the anatomical axis.
* Subjects who have morbid obesity i.e. BMI ≥40.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2004-10; Primary Completion 2010-02 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Number of patients with a functionally stable knee that can achieve post-operative range of motion of 125° or greater. | 1 year
  Proportion of cases that have a functionally stable knee (Q10 of Oxford Knee Score is 'rarely/never' or 'sometimes, or just at first'), AND can achieve 1-year post-op passive range of motion of 125 degrees or greater.

SECONDARY OUTCOMES:
Survivorship of the P.F.C.® Sigma RPF knee at 1, 2, 3, 5, 10, 15 and 20 years. | 1, 2, 3 and 5 years
American Knee Society Change from Baseline Knee and Function Scores at 1, 2, 3, 5, 10, 15 and 20 years | 1, 2, 3 and 5 years
Radiographic assessments at 1, 2, 3, 5, 10, 15 and 20 years | 1, 2, 3 and 5 years
Oxford Knee Score at 1, 2, 3, 5, 10, 15 and 20 years | 1, 2, 3 and 5 years
Patellar Score at 1, 2, 3, 5, 10, 15 and 20 years | 1, 2, 3 and 5 years
SF-12 1, 2, 3, 5, 10, 15 and 20 years | 1, 2, 3 and 5 years

CONTACTS AND LOCATIONS:
Locations (8):
- The Nook, 51/B SV Road, Mumbai, Maharashtra, India
- Kobe University Graduate School Of Medicine, 7-5-1 Kusundki- cho, Chūōku, Kobe, Japan
- Wellington School Of Medicine Surgical Research Trust, Main Street, Newtown, Wellington Region, New Zealand
- Tan Tock Seng Hospital, No 11 Jalan, Tan Tock Seng, Singapore
- Kyunghee University Hospital, 1 HoegiDong, Dongdaemun Gu, Seoul, South Korea
- Sirriraj Hospital, Mahidol University, Bangkok, Thailand
- United Kingdom (2):
  - Nottingham City Hospital, Hucknell Road, Nottingham
  - Clifton Park NHS Treatment Centre, Blue Beck Drive, Shipton Road, York